CLINICAL TRIAL: NCT02816671
Title: MicroCutter Assisted Thoracic Surgery Hemostasis Registry
Acronym: MATCH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AesDex, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-2016-01
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Lobectomy; Segmentectomy
MeSH Terms: interventions — Surgical Staplers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Surgical Stapler — Patients in whom the MicroCutter stapler was used during a thoracic surgical procedure.
  Other Names: MicroCutter Stapler and Reloads

SUMMARY:
The primary purpose of this prospective, open-label, multi-center observational registry with all-comers enrollment is to report on the use of the MicroCutter Stapler in a real world setting in thoracic surgical procedures. Procedures may be open or video assisted thoracic surgery (VATS) including robotic surgical cases. Clinicians will provide objective and subjective evaluation of the use of the stapler in their procedures.

DETAILED DESCRIPTION:
The MATCH registry is a prospective, open label, multi-center observational registry with enrollment of patients requiring surgical stapling during a lobectomy or segmentectomy. Patients will be treated per the clinicians standard of care with medical history and demographic data collected pre-procedure, operative data including clinician's objective and subjective evaluation of the stapler and confirmation of any complications via query and data collection at hospital discharge and each clinician's standard post-operative contact.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lobectomy/segmentectomy in which the MicroCutter Stapler and Reloads were used.
* Patient is willing and able to sign informed consent form to participate in registry, allowing for collection of data.

Exclusion Criteria:

* Clinician determines no vessels are suitable for the on label use of the MicroCutter Stapler and Reloads.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for thoracic surgical procedures requiring the use of a surgical stapler.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2017-11-30 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Hemostasis of vessel staple line | through study completion, approximately 1 month
  Objective classification of hemostasis achieved by the MicroCutter Stapler used on label using a Likert like scale; from 1 (no bleeding) to 5 (bleeding requiring conversion to open procedure or discovered post operatively)

CONTACTS AND LOCATIONS:
Overall Officials: Shanda Blackmon, MD, Principal Investigator — Mayo Clinic; Joel Dunning, PhD, Principal Investigator — James Cook University Hospital
Locations (1):
- James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No